CLINICAL TRIAL: NCT07071363
Title: COMPARATIVE EVALUATION OF THE DERMATOLOGICAL TOLERANCE AND EFFICACY OF A COSMETIC SERUM VERSUS A 4% HYDROQUINONE-BASED PRODUCT IN SUBJECTS WITH MELASMA, AFTER 84 DAYS OF USE - STUDY CONDUCTED UNDER DERMATOLOGICAL SUPERVISION
Brief Title: COMPARISON OF A COSMETIC SERUM AND 4% HYDROQUINONE FOR TREATING MELASMA OVER 84 DAYS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire Dermatologique ACM (Industry)
Collaborators: CIDP Mauritius (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2425CMCL065
Record Dates: First submitted 2025-06-27; First posted 2025-07-17 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Healthy; Melasma (Facial Melasma); Epidermal Melasma
Keywords: Melasma; Hyperpigmentation Skin; Pigmentation Disorders
MeSH Terms: conditions — Melanosis; Hyperpigmentation; Pigmentation Disorders | interventions — hydroquinone

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, controlled, parallel-group study in which subjects are allocated in a 1:1 ratio to one of two intervention arms for a duration of 84 days.
  Group 1 (Cosmetic Product Group): Participants apply Depiwhite Serum (intensive anti-spot serum) in the morning followed by Depiwhite M SPF50+ cream and again apply Depiwhite Serum in the evening followed by a placebo cream (free of hydroquinone).
  Group 2 (Hydroquinone Group): Participants apply a placebo serum (lacking active depigmenting ingredients) in the morning followed by Depiwhite M SPF50+ cream and again apply the placebo serum in the evening followed by Eldopinone cream containing Hydroquinone 4% (USP).
  Both groups follow this regimen for 84 consecutive days. The primary aim is to compare the effectiveness and dermatological tolerance of the cosmetic product versus hydroquinone in subjects with facial melasma.
Who Masked: Participant, Investigator
Masking Description: Investigator is: The principal investigator who was masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depiwhite Serum + Placebo Cream (Experimental): Subjects apply Depiwhite Serum (morning and evening) with Depiwhite M SPF50+ cream in the morning and a placebo cream (no hydroquinone) in the evening for 84 days.
  Interventions: Drug: Depigmenting Cosmetic Serum (Applied Morning and Evening)
- Placebo Serum + Hydroquinone 4% Cream (Active Comparator): Subjects apply a placebo serum (morning and evening) with Depiwhite M SPF50+ cream in the morning and hydroquinone 4% cream (Eldopinone) in the evening for 84 days.
  Interventions: Drug: Depigmenting Cosmetic Serum (Applied Morning and Evening)

INTERVENTIONS:
Drug: Depigmenting Cosmetic Serum (Applied Morning and Evening) — Participants in Group 1 receive a depigmenting cosmetic serum with non-drug actives applied morning and evening, plus a placebo cream without hydroquinone applied in the evening. Group 2 receives a placebo serum (no active depigmenting ingredients) applied morning and evening, and a hydroquinone 4% cream applied in the evening. All participants apply an SPF50+ sunscreen in the morning throughout the 84-day study. The cosmetic serum is the investigational product; hydroquinone serves as the active comparator. Placebo products are visually matched to their respective actives to ensure blinding. The study distinguishes each intervention by active ingredients, timing of application (morning/evening), and role (test vs. reference vs. supportive care). All products are applied topically, and the regimen remains fixed across the study duration.
  Other Names: Hydroquinone 4% Cream (Applied in the Evening); Placebo Serum (Applied Morning and Evening); Placebo Cream (No Hydroquinone, Applied in the Evening); SPF50+ Sunscreen (Applied in the Morning)

SUMMARY:
The goal of this clinical trial is to compare the dermatological tolerance and skin-lightening efficacy of a cosmetic depigmenting serum to a 4% hydroquinone-based product in adult male and female subjects aged 18-65 years with mild to moderate epidermal or mixed-type melasma.

The main questions it aims to answer are:

Does the cosmetic serum reduce the severity of melasma (measured by mMASI) after 84 days of use?

Is the cosmetic serum better tolerated than 4% hydroquinone under real-use conditions?

Researchers will compare the serum group and the hydroquinone group to determine whether the cosmetic product achieves comparable pigmentation improvement with superior skin tolerability.

Participants will:

Group 1: Apply a morning routine (Depiwhite Serum + Depiwhite M SPF50+ cream) Apply an evening routine (Depiwhite Serum + Placebo Cream without Hydroquinone)

Group 2: Apply a morning routine (Serum Placebo + Depiwhite M SPF50+ cream) Apply an evening routine (Serum Placebo + Depigmenting Cream with hydroquinone 4%)

Visit the clinical site at baseline (Day 0), Day 56, and Day 84 for assessments

Complete standardized photographs, self-assessment questionnaires, and quality-of-life surveys (MELASQoL and ASLQI)

Undergo clinical evaluations by a dermatologist, including mMASI scoring and tolerance assessment

DETAILED DESCRIPTION:
Melasma is a chronic hyperpigmentation disorder of multifactorial origin, often aggravated by ultraviolet (UV) radiation, hormonal changes, and inflammation. It predominantly affects individuals with Fitzpatrick skin phototypes III to V and manifests as irregular brown macules and patches, particularly on sun-exposed facial areas. While 4% hydroquinone remains the gold standard topical agent for melasma, its long-term use is associated with adverse events such as irritant dermatitis and exogenous ochronosis, prompting the development of alternative dermocosmetic formulations.

This double-blind, randomized, controlled trial investigates the comparative efficacy and cutaneous tolerance of an intensive anti-spot cosmetic serum (Depiwhite Serum) versus a hydroquinone 4% cream (Eldopinone), both used in conjunction with a high-protection SPF50+ sunscreen (Depiwhite.M). The serum incorporates a combination of active ingredients designed to target melanogenesis and its upstream mediators through a multi-pathway mechanism, including anti-inflammatory, antioxidant, and melanin-regulatory actions.

The study will evaluate changes in melasma severity using a modified Melasma Area and Severity Index (mMASI) score and standardized facial photography acquired with the ColorFace® imaging system. These photographs will undergo high-resolution colorimetric analysis by QIMA Life Sciences, quantifying pigmentation changes through CIELab parameters (L*, a*, b*), ITA°, and contrast metrics (ΔE76, ΔITA°, etc.), tracked across predefined regions of interest (ROIs) from lesional and perilesional skin.

Additional assessments include subjective product performance evaluation, cosmetic acceptability, and patient-reported outcomes using two validated quality-of-life instruments (MELASQoL and ASLQI). Safety and local tolerance will be monitored at each clinical visit via dermatologist-led skin examinations and subject-reported functional symptoms.

The trial aims to generate robust clinical and instrumental data supporting the use of cosmetic formulations as a potential alternative or maintenance therapy to hydroquinone in melasma management, particularly for populations seeking better tolerability profiles without compromising efficacy.

Amendment Note (15 August 2025 The inclusion criteria have been revised to allow subjects with a baseline mMASI score of ≥3.5 (previously ≥4) to accommodate borderline moderate melasma cases. This change is reflected in Protocol Version 2.0.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects, primarily female, aged 18 to 65 years at the time of inclusion

Fitzpatrick skin phototype II to V

Diagnosed with mild to moderate epidermal or mixed-type facial melasma, confirmed by Wood's lamp examination

mMASI score between 3.5 and 13 at baseline

Subject is in general good health as assessed by the investigator based on medical history and clinical examination

Willing to avoid excessive sun exposure and use only the provided SPF50+ sunscreen during the study

Able to understand the study procedures and provide written informed consent

Willing and able to comply with study procedures and scheduled visits

Women of childbearing potential must agree to use a reliable method of contraception for at least 3 months prior to and during the entire study duration

Exclusion Criteria:

Presence of post-inflammatory hyperpigmentation (PIH), lentigines, or other non-melasma facial pigmentation

Use of topical or systemic depigmenting treatments, retinoids, corticosteroids, or hormonal treatments within 4 weeks prior to baseline

Known allergy or hypersensitivity to any component of the investigational or comparator products

Excessive sun exposure or use of tanning beds within 2 weeks before baseline or planned during the study

Active skin diseases (e.g., atopic dermatitis, psoriasis) or damaged skin in the test area

Pregnant or breastfeeding women, or those planning to become pregnant during the study

Participation in another clinical trial within 4 weeks prior to the study or planned participation in another trial during the study

History of malignancy in the past 10 years (except treated basal cell carcinoma)

Uncontrolled systemic illness (e.g., diabetes, cardiovascular, hepatic, renal, or pulmonary disease)

Any psychological or cognitive condition that would limit the subject's ability to understand the study procedures

Current use of photosensitizing medications

BMI > 40 or other conditions that may affect protocol compliance as judged by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Melasma Area and Severity Index (mMASI) Score From Baseline (Day 0) to Day 84 ±1 Day, Assessed by a Blinded Dermatologist to Evaluate the Clinical Efficacy of the Investigational and Comparator Products in Subjects With Melasma | Baseline (Day 0) to Day 84 ±1 day. The mMASI score will be assessed at both time points by a blinded dermatologist to evaluate the change in melasma severity over the 12-week treatment period.
  The modified Melasma Area and Severity Index (mMASI) is a validated clinical scoring method used to assess the severity and extent of facial melasma. It evaluates four facial regions (forehead, right malar, left malar, and chin) based on the area of involvement and the intensity of pigmentation. Each region contributes proportionally to the total score, which ranges from 0 (no melasma) to 24 (severe melasma). In this study, the mMASI score will be assessed by a blinded dermatologist at baseline (Day 0) and again at Day 84 (±1 day). The primary objective is to quantify the change in mMASI score after 12 weeks of treatment with either the investigational cosmetic serum (Depiwhite Serum) or the comparator product containing hydroquinone 4% (Eldopinone). This outcome will serve as the primary measure of clinical efficacy in reducing melasma severity over the course of the study.

SECONDARY OUTCOMES:
Change in modified Melasma Area Severity Index (mMASI) at Day 56 | Day 56
  Clinical evaluation of melasma severity on each hemi-face using the modified mMASI score, comparing baseline to Day 56.
  Unit of measure: Score(0-24)
Change in Individual Typology Angle (ITA°) from baseline | Day 56 and Day 84
  Evaluation of melasma pigmentation using ITA° from standardized ColorFace® photographs. Two Regions of Interest (ROI) are analyzed: one in melasma-affected skin and one in adjacent healthy skin.
  Unit of Measure: Degrees (°)
Change in Melasma Quality of Life Index (MELASQoL) | Day 56 and Day 84
  Subjects complete the MELASQoL questionnaire to evaluate the emotional and social impact of melasma.
  Unit of Measure: Score (7-70)
Subject-rated product efficacy and cosmetic acceptability | Day 28, Day 56, and Day 84
  Subjects assess perceived product performance (e.g., brightness, evenness, spot reduction) and cosmetic acceptability using a structured questionnaire.
  Unit of Measure: Score on 4-point scale
Investigator-assessed dermatological tolerance | Day 56 and Day 84
  Evaluation of local intolerance signs (e.g., erythema, dryness, desquamation) by dermatologist using a standardized clinical scale.
  Unit of Measure: Severity score (0-4 scale)
Subject-reported local intolerance symptoms | Day 56 and Day 84
  Description: Subjects report symptoms such as burning, itching, stinging, and tightness on the face using a self-assessment scale.
  Unit of Measure: Severity score (0-4 scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre International de Développement Pharmaceutique, Port Louis, Phoenix, Mauritius

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared for this study. The trial involves cosmetic products and is not subject to regulatory requirements mandating data sharing. Additionally, participant privacy and confidentiality are prioritized, and the data collected are not intended for secondary research use.